CLINICAL TRIAL: NCT00155467
Title: Establish a CT Images Database of Patients With Congenital Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9461700815
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-10-20 (Estimated); Status verified 1995-01

CONDITIONS: Heart Diseases
Keywords: CT; children; congenital
MeSH Terms: conditions — Heart Diseases

INTERVENTIONS:
Procedure: CT

SUMMARY:
Setup CT images database of congenital heart disease.

DETAILED DESCRIPTION:
Setup CT images database of congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

- congenital heart disease

Exclusion Criteria:

-

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5000
Dates: Start 1995-01; Study Completion 2010-12

PRIMARY OUTCOMES:
diagnostic accuracy

SECONDARY OUTCOMES:
senstivity
specificity

CONTACTS AND LOCATIONS:
Overall Officials: Shyh-Jye Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Dept. Medical Imaging, NTUH, Taipei, Taiwan